CLINICAL TRIAL: NCT05940129
Title: Integrating Maternal, Fetal, Newborn or Infant Safety in Antenatal and Post-natal Care Services for Rural and Tribal Women in India
Brief Title: Women and Child, Safety, Health, and Empowerment
Acronym: WC-SHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00278599
Record Dates: First submitted 2023-06-28; First posted 2023-07-11 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Gender-based Violence
MeSH Terms: interventions — Safety; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Web-based Intervention Arm (WC-SHE) (Experimental): Women in computerized WC-SHE arm receives education on healthy relationships the danger assessment and tailored safety planning and list of resources. The intervention also includes assessments of strengths and safety strategies. In addition, husbands and in-laws receive one-on-one health education session that includes topics related to maternal and child health and safety
  Interventions: Behavioral: Women and Child, Safety, Health and Empowerment (WC-SHE)
- WC-SHE +Economic Empowerment (Experimental): Women in economic empowerment arm receive computerized WC-SHE and are connected with self-help groups. Husbands are also engaged in economic empowerment activities that involve individual psychoeducation, working with spouses in self-help group activities and participating in government economic or vocational training programs. In addition, husbands and in-laws participate in individual sessions on topics related to maternal and child health and safety
  Interventions: Behavioral: Women and Child, Safety, Health and Empowerment (WC-SHE)
- WC-SHE + Enhanced Family Psychoeducation and Advocacy Support Intervention (Experimental): Women in this arm receive computerized WC-SHE, advocacy and support by a support committee of professionals based on women's priorities and needs, and phone call support by women community resource persons. Husbands and in-laws participate in individual and group sessions that cover topics such as stress, healthy relationships, healthy communication within families and impact of domestic violence on children.
  Interventions: Behavioral: Women and Child, Safety, Health and Empowerment (WC-SHE)

INTERVENTIONS:
Behavioral: Women and Child, Safety, Health and Empowerment (WC-SHE) — The WC-SHE component includes a risk assessment and tailored safety planning for women in domestic violence relationships. In addition, the component involves one-on-one education with husbands and in-laws. The economic empowerment component is designed to support women and their husbands in economic empowerment activities. The advocacy arm involves community education of husbands and in-laws, advocacy support by a support committee comprised of multidisciplinary professionals and phone support by women community resource persons

SUMMARY:
Gender-based violence (GBV) (including homicide) is one of the leading causes of maternal and child (fetus, newborn or infant) mortality and morbidity in limited resource settings such as India. This study is evaluating the feasibility, acceptability and preliminary efficacy of WC-SHE (Women and Children-Safety, Health and Empowerment) intervention developed to promote health and safety outcomes of mother and children in rural and/or tribal regions in India. The aim will be to refine, optimize and standardize the WC-SHE intervention and its added components, develop fidelity measures, conduct a feasibility and acceptability evaluation of the intervention and implementation procedures as well as examine preliminary efficacy outcomes of WC-SHE.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years of age
2. Currently pregnant
3. Experienced intimate partner and/or in-law abuse in the past
4. Residing in rural or tribal areas in India

Exclusion Criteria:

1. Under 18 years of age
2. Not currently pregnant
3. No experience of intimate partner and/or in law abuse
4. Not residing in rural or tribal areas in India

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 150 (Actual)
Dates: Start 2022-10-21 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Severity and frequency of abuse by husband and in-laws as measured by the adapted Conflict Tactics Scale (CTS2) | Baseline, 3 months, 6 months
  Severity and frequency of abuse is assessed by the adapted version of the Revised Conflict Tactics Scale . Response categories range from 0 (never) to very 7 (frequently). Higher overall scores mean more conflict. Measured at Baseline, 3 months, 6 months.
Number of maternal safety behaviors as assessed by the Safety Behavior Checklist | Baseline, 3 months, 6 months
  The Safety Behavior Checklist is used to measure the number of safety strategies and support services used. Measured at Baseline, 3 months, 6 months.
Victim empowerment related to safety as assessed by the Measure of Victim Empowerment Related to Safety (MOVERS) Scale | Baseline, 3 months, 6 months
  The MOVERS scale is a 13 item scale that measures survivor empowerment within the domain of safety. Participants respond to each item using a five-point Likert scale (from "never true" to "always true. Possible score range 13-65. Higher scores indicate higher levels of empowerment related to safety. Measured at Baseline, 3 months, 6 months.
Uncertainty in choosing safety options as assessed by the Adapted Decisional Conflict scale | Baseline, 3 months, 6 months
  The Adapted decisional conflict scale is used to measure decisional conflict for safety. The response options ranged from strongly disagree to strongly agree, with higher scores indicating lower decisional conflict. Decisional Conflict Scale scores range from 0(no decisional conflict) to 100 (high decisional conflict). Measured at Baseline, 3 months, 6 months.
Depression as assessed by the Patient Health Questionnaire | Baseline, 3 months, 6 months
  The Patient Health Questionnaire (PHQ-9) is used to measure depression; Total scores of 5, 10, 15, and 20 represent cut points for mild, moderate, moderately severe and severe depression. Score range 0-27. Measured at Baseline, 3 months, 6 months.
Probable Post Traumatic Stress Disorder (PTSD) in primary care settings | Baseline, 3 months, 6 months
  Primary Care PTSD Screen is a 5 item screen used to identify participants with probable PTSD in primary care settings. The items are rated on a binary scale (No, Yes). Score range 1-5. Higher scores indicate increased post traumatic stress symptoms. Measured at Baseline, 3 months, 6 months.
Physical health status | Baseline, 3 months, 6 months
  For self-rated physical health, participants are asked about how would they describe their health during pregnancy (or post-delivery). The response options include poor, fair and excellent with poor coded as 1, fair as 2 and excellent as 3. Measured at Baseline, 3 months, 6 months.
Fetal safety as measured by occurrence of fetal loss | Post intervention up to 6 months
  Fetal loss includes post-intervention occurrence of any induced abortion or miscarriage, spontaneous abortion or miscarriage, or occurrence of fetal mortality or still birth
Newborn/infant safety as measured by self-reported items developed by the study team | 6 months
  The following items are used to measure newborn or infant safety, (a) participants are asked about concern for the child's mistreatment by the participants husband or in-laws. The response options range from never (0) to always (4). (b) Participants are asked if there is concern about harm to the child by anyone, with yes/no response options; Any incident of death of a child within few weeks post-delivery is based on participants' self-reports
Newborn/infant health as measured by two items developed by the study team | 6 months
  Newborn/infant health is measured by number of participants who delivered a low birth weight or pre-term child. Participants are asked if newborn was (a) a low birthweight child; and (b) child born preterm.
Level of satisfaction with child's health and health-related issues as assessed by the Postpartum Quality of Life (PQOL) measure | 6 months
  Participants are asked adapted items from the child care dimension of the Postpartum Quality of Life (PQOL) measure. The response options for items range from very dissatisfied to very satisfied and frequency levels ranging from never to always. Score range 16-80, with higher scores showing better quality of life.

SECONDARY OUTCOMES:
Self-efficacy for safety as assessed by an item developed by study team | Baseline, 3 months, 6 months
  Self-efficacy for safety is measured using one item that assesses for the level of confidence women have in their ability to implement measures to keep themselves safe from experiencing abuse and mistreatment. The response options range from not confident at all to very confident. Measured at Baseline, 3 months, 6 months.
Resilience as assessed by the Connor Davidson Resilience Scale | Baseline, 3 and 6 months
  Resilience is measured using the 10-item Connor-Davidson Resilience Scale; Respondents rate items on a 5-point Likert scale, ranging from 0 (not true at all) to 4 (true nearly all the time). Each item has a minimum score of 0 and a maximum score of 4.
Sources of support as assessed by the Brief Perceived Social Support Questionnaire | Baseline, 3 months, 6 months
  Perceived sources of support are measured using the Brief Perceived Social Support. The questionnaire.measures general perceived social support with a 6 item, five-point Likert scale ranging from 1 (not true at all) to 5 (very true). Higher scores indicate higher levels of perceived social support. Possible score 6-30. Measured at Baseline, 3 months, 6 months.
Number of Self- care behaviors as measured by the items developed by the study team | Baseline, 3 months, 6 months
  Women are asked about the number of care visits and visits to healthcare providers for specific health concerns. Change in self care behaviors will be assessed by change in attending the minimum number of recommended care visits; and number of visits to medical providers for health concerns. Measured at Baseline, 3 months, 6 months.
Economic stress | Baseline, 3 months, 6 months
  Participants are asked about how often they ran out of money for necessities (e.g., food, housing etc for themselves or/and their children). The response options include never, once or twice, every month or monthly, every week or weekly, every day or daily. Measured at Baseline, 3 months, 6 months.
  .

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Sabri, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No